CLINICAL TRIAL: NCT00747539
Title: Neurobehavioral Deficits in HIV/HCV Infection Pre/Post Anti-HCV Therapy
Brief Title: Brain Deficits in HIV/HCV Coinfected People Before and After Anti-HCV Therapy
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Charles Hinkin, Ph.D, University of California, Los Angeles
Other Study IDs: R01MH083553 (NIH); R01MH083553 (NIH); DAHBR 9A-ASNM
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: HIV; Hepatitis C; Infections
Keywords: Hepatitis C Virus; HCV; Human Immunodeficiency Virus; Coinfection
MeSH Terms: conditions — Hepatitis C; Infections; Acquired Immunodeficiency Syndrome; Coinfection | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: This group will be composed of 165 HCV-infected people who are not also HIV infected.
  Interventions: Drug: Pegylated interferon alfa and ribavirin (PEG-IFN/RBV)
- 2: This group will be composed of 165 HCV-infected people who are also HIV infected.
  Interventions: Drug: Pegylated interferon alfa and ribavirin (PEG-IFN/RBV)

INTERVENTIONS:
Drug: Pegylated interferon alfa and ribavirin (PEG-IFN/RBV) — Pegylated interferon alfa and ribavirin (PEG-IFN/RBV), considered standard care for patients with chronic HCV, will be given to participants.
  Other Names: Pegasys

SUMMARY:
This study will evaluate the impact of standard hepatitis C virus treatment on brain deficits in people who are infected with both HIV and the hepatitis C virus.

DETAILED DESCRIPTION:
The World Health Organization estimates at least 3% of the world's population is infected with chronic hepatitis C virus (HCV), and up to one third of all HIV infected people are coinfected with HCV. HCV can damage the liver cells and cause liver diseases such as cirrhosis and hepatocellular carcinoma. People infected with HCV can also suffer from neurocognitive deficits, including problems with information processing, slowing of muscular processes related to thinking, and difficulty focusing on complex things. These neurocognitive deficits are similar to those found in HIV infected individuals, and previous research indicates that people infected with both HIV and HCV have greater overall cognitive impairments. This study aims to determine the impact of anti-HCV treatment on neurocognitive, neuropsychiatric, and neuroimaging factors in people infected with HCV and people coinfected with both HCV and HIV. The study also aims to measure whether possible neurocognitive improvements from anti-HCV treatment are related to a physical health outcome, measured as a sustained virologic response, and whether adherence to the medication schedule laid out for the participants influences possible positive effects on either neurocognitive or physical health.

Two kinds of participants will be recruited for this study: those infected with HCV and those infected with both HCV and HIV. These two groups will be compared to determine how comorbid HCV and HIV infection affects treatment outcomes. The treatment specified for HCV is pegylated interferon alfa and ribavirin (PEG-IFN/RBV), considered standard care for patients with chronic HCV. Participants will continue to see their doctors as regularly scheduled, and any other prescribed medications or advice concerning HCV treatment will be noted by researchers. All participants will be tested at baseline, after 12 weeks of treatment, and 12 weeks after the completion of treatment. A subset from each group of participants will undergo additional neuroimaging tests. Participation in this study will last for varied amounts of time depending on the recommended treatments for HCV. Based on each virus' genotype and rapid virologic response, the treatment period for HCV may last 24 or 48 weeks, with further extensions of 12 to 24 weeks in some cases.

During the three testing sessions, each lasting 5 hours, participants' health, cognitive functioning, and medication adherence will be measured. Testing will include self-report measures, intelligence tests, tasks designed to assess cognitive functioning, and motor functioning tasks. Urine tests screening for narcotics will also be collected. In addition to self-report measures, caps to pill bottles storing HCV medication will automatically record every time the cap is removed to measure adherence to the medication schedule.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCV with detectable HCV RNA in serum
* Meets clinical criteria for initiating HCV therapy
* Lives in the community and not in a board and care, nursing home, hospice, or other residential setting in which a professional caregiver would dispense necessary medication. Living with a partner, roommate, or other family members who may assist with caregiving, including reminding participants to take medication, is acceptable.
* Responsible for administering own medications
* Diagnosis of HIV-associated neurocognitive disorder (HAND) will not be cause for exclusion, so long as participant is able to demonstrate the ability to grant full informed consent
* HIV or HCV disease severity will not be cause for exclusion (e.g., CDC Groups A, B, and C are all eligible); although, if severely ill because of either HIV (e.g., uncontrolled viremia, severely immunosuppressed) or HCV (e.g., cryoglobulinemia, hepatic encephalopathy) will not be eligible for PEG-IFN/RBV therapy
* Able to read English at the 6th grade level

Exclusion Criteria:

* Current or past psychotic spectrum disorder, including schizophrenia, schizophreniform disorder, or bipolar disorder
* History of learning disability, seizure disorder, closed-head injury with loss of consciousness in excess of 30 minutes, or any other neurological disease
* Evidence of any central nervous system opportunistic infection or neoplasm
* Diagnosed with Hepatitis B
* Previous failed course of HCV therapy
* Those judged to be significantly depressed by the study psychiatrists/psychologists (defined as current major depressive disorder of moderate or severe severity) or with evidence of suicidal ideation will not be enrolled until clinical condition is stabilized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 165 HCV-monoinfected and 165 HIV/HCV-coinfected participants who are receiving HIV and/or HCV treatment through the VA Greater Los Angeles Health Care System, the AIDS Healthcare Foundation, or the Kaiser-Permanente Infectious Disease Program.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2008-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral deficits as observed on neuropsychological testing in HIV/HCV-coinfected individuals before and after receiving anti-HCV treatment. | Measured before drug administration, Week 12 of drug administration, and Week 12 of follow-up

SECONDARY OUTCOMES:
Psychiatric symptoms | Measured before drug administration, Week 12 of drug administration, and Week 12 of follow-up
Neuroimaging data (from a nested cohort of participants) | Measured before drug administration, Week 12 of drug administration, and Week 12 of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Charles H. Hinkin, PhD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - Kaiser Permanente Infectious Diseases, Antelope Valley, Lancaster, California
  - University of California, Los Angeles, School of Medicine, Los Angeles, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Veterans Administration Greater Los Angeles Healthcare System, Los Angeles, California